CLINICAL TRIAL: NCT06933433
Title: A Retrospective Analysis of Assaults Against Health Care Professionals in a Tertiary Intensive Care Unit
Brief Title: Assaults Against Health Care Professionals in a Tertiary Intensive Care Unit
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2024-00927; am25Sutter
Record Dates: First submitted 2025-03-25; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Assault
Keywords: Workplace violence; Intensive care unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the occurrence of workplace violence, both physical, verbal, and sexual assaults, from patients and their relatives towards intensive care unit staff members.

DETAILED DESCRIPTION:
Workplace violence, as defined by the International Labor Organization, includes any action, incident, or behavior that assaults, threatens, harms, or injures a person during their work. Healthcare workers face the highest risk of workplace violence among all professions. Violence can take many forms, including verbal abuse, physical offenses to sexual harassment. While most research focuses on psychiatric and emergency departments, workplace violence in intensive care units (ICUs) is understudied and often underreported.

As a result, little is known about its prevalence and risk factors, leading to a lack of awareness and effective prevention strategies. The aim of this retrospective single-center cohort study is to investigate the occurrence of workplace violence, both physical, verbal, and sexual assaults, from patients and their relatives towards ICU staff members. The study will assess the frequency, characteristics, and circumstances of these events in an intensive care setting. Additionally, the consequences of such incidents and the measures taken afterward will be examined. This analysis aims to identify potential risk factors and possible targets for intervention, ultimately contributing to the development and implementation of protocols that enhance the safety of both healthcare professionals and patients.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Reported incident of physical, verbal or sexual violence in the intensive care unit at the University Hospital Basel

Exclusion Criteria:

None defined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive adult patients (i.e.≥ 18 years of age) with a reported incident of physical, verbal or sexual violence in the intensive care unit at the University Hospital Basel from January 1st 2011 until end of June 2024 as documented in the digital medical records.
Sampling Method: Probability Sample
Enrollment: 865 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Demographic information | 2011-06/2024
  Demographic information of persons involved in the assault (e.g., age, sex, function) is collected.
Acute prehospital management data | 2011-06/2024
  Data from acute prehospital management, as documented in emergency medical services (EMS) treatment protocols, is collected. The collected data elements are aggregated to describe the overall EMS response.
Duration of intensive care unit stay | 2011-06/2024
  The length of intensive care unit (ICU) stay is recorded.
Duration of hospital stay | 2011-06/2024
  The length of the total hospital stay is recorded.
Discharge destination | 2011-06/2024
  The destination at discharge (e.g., other hospital, nursing home, hospice, rehabilitation, or home) is recorded .
Date of assault | 2011-06/2024
  The specific date of reported workplace violence is documented.
Characteristics of assault | 2011-06/2024
  Details on the assault incident as documented in nurses' and physicians' progress notes (e.g. wording) to characterize the event.
Type of assault | 2011-06/2024
  The type of workplace violence (e.g. verbal, physical, emotional) is recorded.
Additional features of the assault | 2011-06/2024
  Assessment of additional features related to workplace violence, including involved staff members, shift type, and environment. These features are aggregated to characterize the context in which the assault occurred.
Patient characteristics | 2011-06/2024
  Information on the patient (e.g., main diagnosis, comorbidities, medication) is documented.
Consequences of the assault | 2011-06/2024
  Evaluation of the consequences, including staff changes, safety measures, and debriefing following workplace violence incidents.
Neurological status based on validated clinical assessment | 2011-06/2024
  Neurological status during ICU stay is assessed using available data in the patient register from validated neurological assessments. These may include the Richmond Agitation-Sedation Scale (RASS), Sedation-Agitation Scale (SAS), Glasgow Coma Scale (GCS), Intensive Care Delirium Screening Checklist (ICDSC), or Status Epilepticus Severity Score (STESS). The specific tool used, as well as the scale of the score and meaning behind the score, depends on routine clinical practice and available documentation in the register. If multiple scores are available for a patient, they will be aggregated to provide a comprehensive assessment of neurological status.
Critical illness severity score | 2011-06/2024
  Disease severity is assessed using standardized scoring systems, such as Acute Physiology and Chronic Health Evaluation II (APACHE II), Simplified Acute Physiology Score II (SAPS II), and Sequential Organ Failure Assessment (SOFA) scores. The scale of the score and meaning behind the score depends on the severity assessment that is applied.
Charlson Comorbidity Index | 2011-06/2024
  The Charlson Comorbidity Index (CCI) is calculated based on pre-existing comorbidities and additional diagnoses. The CCI predicts the ten-year mortality for a patient who may have a range of comorbid conditions. It assigns weighted scores (from 0 to maximal 6) to 17 comorbid conditions (e.g., heart disease, diabetes, cancer), resulting in a total score ranging from 0 to 33, if the patient had the most severe form of each of the 17 conditions.
Laboratory parameters | 2011-06/2024
  Routine laboratory value for e.g. C-Reactive Protein (CRP), albumin, Lactate Dehydrogenase (LDH), Creatine Kinase (CK), procalcitonin, white blood cell levels, creatinine, liver enzymes, blood gas analyses, and metabolic data, is collected. The specific parameters recorded may vary depending on the laboratory assessments documented in the patient register. All values will be reported using their respective units of measurement.
Glasgow Outcome Score | 2011-06/2024
  The Glasgow Outcome Score (GOS) is calculated based on the assessment of key clinical outcomes such as in-hospital mortality, survival, survival with neurofunctional alteration, return to premorbid neurological function, and hospital readmission to determine the patient outcome.
  The GOS ranges from 1 (death) to 5 (good recovery).
Therapeutic intervention | 2011-06/2024
  The therapeutic intervention is document, including information on duration, dosage and number of treatment medication, number of neuroleptic, sedative and analgesic drugs, invasive procedures, such as intubation, mechanical, ventilation, vasopressors, installation of central lines, nutrition, etc.
Vital signs | 2011-06/2024
  Vital signs are analyzed based on the data available in the patient register. These may include blood pressure, heart rate, respiratory rate, oxygen saturation, body temperature, and level of consciousness. The specific parameters recorded depend on the clinical documentation available. All values will be reported using their respective units of measurement. The collected parameters are aggregated to provide an overall assessment of the patient's clinical condition.
Fluid balance data | 2011-06/2024
  Fluid balance data, including the administration of fluids such as blood products, crystalloids, and enteral/parenteral nutrition, are documented. These components are aggregated to represent overall fluid input for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Raoul Sutter, Prof. Dr. med., Principal Investigator — University Hospital Basel, Department of Acute Medicine, Intensive Care Unit
Locations (1):
- University Hospital Base, Intensive Care Unit, Basel, Canton of Basel-City, Switzerland